CLINICAL TRIAL: NCT03979001
Title: Pilot Study: Retinal Vascular Network and Obstructive Sleep Apnea
Brief Title: Retinal Vascular Network and Obstructive Sleep Apnea
Acronym: ORNET
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GABRIELLE 2018
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients referred for polysomnography diagnosis of obstructive sleep apnea syndrome
  Interventions: Other: complete ophthalmological examination
- Controls: Person without obstructive sleep apnea syndrome

INTERVENTIONS:
Other: complete ophthalmological examination — collection:
  * ophthalmological history and current treatments
  * occular tension measurement
  * measurement of visual acuity (Snellen chart)
  * Axial length measurement
  * Photograph of the posterior segment of the eye
  * 3x3 and 6x6 macular and papillary OCT angiography
  Groups: Patients

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is thought to lead to systemic vascular lesions that may be preceded by early microvascular lesions in the eyes and in particular in the retina. The improvement of ophthalmological imaging techniques by OCTangiography allows a precise non-invasive study of the retinal microvascular network. This new rapid and non-invasive retinal imaging tool could reveal micro-vascular lesions related to OSA. To the investigator's knowledge, this would be the first OCT-angiography description of a cohort of patients with OSA. If these results are confirmed, it would be interesting to study the correlation between these micro-vascular lesions and the cardiovascular risk of his patients.

ELIGIBILITY:
Inclusion Criteria:

* person who has given oral consent
* person who can be followed throughout the study
* adult

Patient group:

- Patient seen in sleep apnea screening consultation by a pulmonologist and referred for polysomnography diagnosis of OSA

Control Group:

- Person initially without obstructive sleep apnea syndrome

Exclusion Criteria:

* a person who is not affiliated to or not a beneficiary of the national health insurance system
* person subject to a measure of legal protection (curatorship, guardianship)
* person subject to a safeguard of justice
* pregnant, parturient or breastfeeding woman
* adult incapable or unable to consent
* person with a contraindication to Tropicamide or Neosynephrine
* person with a history of eye disease affecting ocular circulation (examples: acute anterior ischemic optic neuropathy, retinal central artery occlusion, retinal central vein occlusion, diabetic retinopathy, glaucoma, uncontrolled hypertonia, AMD, severe myopia...)

Control Group:

* person with a history of chronic lung problems (e.g. COPD, chronic respiratory failure, etc.)
* person with at least one of the following risk factors for obstructive sleep apnea syndrome:

  * Obesity with IMC≥30
  * Alcohol consumption > 3 glasses per day

Exclusion criteria: positive result in one of the 3 self-questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen for sleep apnea screening by a pulmonologist and referred for polysomnography diagnosis of obstructive sleep apnea syndrome
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Measurement of macular and peri-papillary retinal vascular density of the superficial and deep capillary plexuses | Change from baseline at 24 months
Measurement of macular and peri-papillary retinal infusion density of the superficial and deep capillary plexuses | Change from baseline at 24 months
Measurement of the surface of the macular avascular zone of the superficial and deep capillary plexuses | Change from baseline at 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No